CLINICAL TRIAL: NCT03949504
Title: Early Diagnosis and Management of Patients at Risk for Diabetes
Brief Title: Diabetes Risk Diagnosis and Management
Acronym: DIARIO
Status: Completed | Type: Observational
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Licia Iacoviello, MD, PhD, Neuromed IRCCS
Other Study IDs: DEP3_2019
Record Dates: First submitted 2019-05-09; First posted 2019-05-14 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; neurological complications; cardiovascular complications
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General population: Male and Female subjects (n=1000) over 34 years of age randomly recruited from the participants to the recall phase of the Moli-sani study
  Interventions: Procedure: New Find-risk questionnaire software
- Patients with type 2 Diabetes: Male and Female patients with type 2 diabetes (n=550) without (n=200) or with cardiovascular (n=200) or neurological (n=150) complications consecutively admitted to the IRCCS Neuromed

INTERVENTIONS:
Procedure: New Find-risk questionnaire software — FINDrisk: software with 12 questions to define the risk of diabetes in the general population MyStar Connect: software to guide the diagnosis and the management of diabetes and its complications
  Other Names: MyStar Connect software (version beta)
  Groups: General population

SUMMARY:
Considering the multifactorial nature of the complications of Type 2 diabetes, such as cardiovascular and neurological complications and therefore the multiplicity of risk factors that contribute to their development, it is assumed that the use of a dedicated function of the MyStar Connect software (beta version), that allows the querying of the application through specific queries (presence of risk factors) and the calculation of specific risk scores in order to extract the patients most at risk of developing such complications, can provide support to the diabetologist to optimize management of the patient at risk and complicated through, for example, a more intensive visit program and this then translates into an improvement in the parameters related to these risk factors.

DETAILED DESCRIPTION:
The study aims are:

* To evaluate the percentage of subjects at risk of diabetes in the general population
* To evaluate the percentage of type 2 diabetics with and without complications in the identified population at risk
* To evaluate whether the new computer system is able to identify subjects at risk of developing complications or aggravation of complications already in progress (cardiovascular and neurological complications).

Through the IT platform made available within the framework of the project, the selected sample will be given the questionnaire to detect the risk of diabetic disease (FINDRISC adapted) and, in the case of a positive outcome, the subject at risk will be assessed with laboratory tests, to confirm or not the condition of prediabetes or diabetes. Therefore, all the subsequent phases of patient care and management will be followed, from the modification of lifestyles for prediabetics to the management of overt diabetic pathology and the complications associated with it, thus experimenting with all the modules of the software platform integrated.

Subjects who have a high diabetic risk score will be referred to the Neuromed laboratories for the analysis of fasting blood glucose and the glycemic load test. Consistent with the diagnostic protocol developed, the subjects will follow a triple address:

1. Subjects at risk with fasting blood glucose or normal glycemic load
2. Subjects with prediabetes
3. Subjects with diabetes Patients in whom a vascular or neurological complication is diagnosed will be managed by the Neuromed clinic work groups using dedicated modules developed within the project.

At time T0 for diabetic patients without or with cardiovascular and neurological complications who will come to visit as from normal clinical practice, the presence of risk / complication parameters will be checked and risk scores will be applied to ascertain the patient's condition. The patient will then be followed as per normal clinical practice and risk parameters and the derived scores will be re-evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Signature of informed consent;
* Subjects recruited consecutively during the recall phase of the Moli-sani project.
* Patients with type 2 diabetes mellitus and vascular or neurological complications attending the IRCCS Neuromed

Exclusion Criteria:

* Inability to understand and to want
* Refusal to sign informed consent.
* Type 1 diabetes
* Gestational diabetes.
* For subjects of the general population, a previous diagnosis of diabetes.

Ages: 34 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive male and female subjects, over 34 years of age recruited in teh framework of the recall phase of the Moli-sani study.
  Male and Female patients with type 2 diabetes without or with cardiovascular or neurological complications
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Number of subjects at high risk for Diabetes | 12 months
  Risk for type 2 diabetes measured by a structured questionnaires with 11 questions scoring from -1 to 27 and classified in 5 risk categories: Low risk (score>6); Low-medium risk (score 7-11); Medium-high risk (score 12-14); high risk (score 15-20); very high risk (score >20).
Number of subjects with diabetes | 18 months
  diabetes diagnosis will be based on fasting plasma glucose (FPG)≥126 mg/dl. The testswill be performed in a laboratory using a certified method. Fasting is defined as no caloric intake for at least 8 h.
Concentration of glucose in plasma | 24 months
  Glucose control in patients with diabetes and cardiovascular or neurological complications, measured with plasma glucose criteria, defined as FPG <126 mg/dL (7.0 mmol/L).

CONTACTS AND LOCATIONS:
Overall Officials: Licia iacoviello, MD, PhD, Principal Investigator — IRCCS Neuromed
Locations (1):
- IRCCS INM Neuromed, Department of Epidemiology and Prevention, Pozzilli, IS, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Result] Lindstrom J, Tuomilehto J. The diabetes risk score: a practical tool to predict type 2 diabetes risk. Diabetes Care. 2003 Mar;26(3):725-31. doi: 10.2337/diacare.26.3.725. PMID 12610029
- [Result] Bergmann A, Li J, Wang L, Schulze J, Bornstein SR, Schwarz PE. A simplified Finnish diabetes risk score to predict type 2 diabetes risk and disease evolution in a German population. Horm Metab Res. 2007 Sep;39(9):677-82. doi: 10.1055/s-2007-985353. PMID 17846976
- [Result] Li J, Bergmann A, Reimann M, Bornstein SR, Schwarz PE. A more simplified Finnish diabetes risk score for opportunistic screening of undiagnosed type 2 diabetes in a German population with a family history of the metabolic syndrome. Horm Metab Res. 2009 Feb;41(2):98-103. doi: 10.1055/s-0028-1087191. Epub 2008 Oct 29. PMID 18975253
- [Result] American Diabetes Association. Diagnosis and classification of diabetes mellitus. Diabetes Care. 2010 Jan;33 Suppl 1(Suppl 1):S62-9. doi: 10.2337/dc10-S062. No abstract available. PMID 20042775